CLINICAL TRIAL: NCT06070155
Title: Effect of Aerobic Exercises on Some Trace Elements and the Quality of Life in Post-menopausal Women After Radiotherapy
Brief Title: Effect of Aerobic Exercises on Trace Elements in Post-menopausal Women After Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tarek Hussein Mostafa, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004581
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Trace Elements Levels After Breast Cancer Radiotherapy
Keywords: trace elements; breast cancer; aerobic exercise
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Aerobic exercises and no intervention
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise three times a week (Experimental): The participants will receive mild to moderate aerobic exercise for three weeks for 12 sessions.
  Interventions: Other: Aerobic Exercise three time a week
- No Exercise group (No Intervention): This group will act as a control group.

INTERVENTIONS:
Other: Aerobic Exercise three time a week — The participants will receive mild to moderate aerobic exercise for three weeks for 12 sessions.
  Arms: Aerobic exercise three times a week

SUMMARY:
This study will be conducted on 28 participants who are survivors of breast cancer and underwent radiotherapy. The purpose of the current study is to investigate the effect of aerobic exercises on quality of life and serum levels of Zinc, Copper and iron in post-menopausal women who received radiotherapy after surviving breast cancer.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common type of cancer in women globally. Several studies observed changes in the serum blood levels of trace elements in BC. Essential trace elements have relevant functions in a large number of cellular processes, with multiple roles in the correct functioning of metabolic enzymes.

There were previous trials to investigate the effect of exercise on trace elements in different populations as in the elite sportsmen. Some other studies to investigate the effect of exercise on breast cancer survivors for instance (Duijts et al., 2011) stated that physical exercise has effects on psychosocial functioning and health-related quality of life in breast cancer patients and survivors. Also, (Lambrigts et al., 2022) stated that aerobic exercise is the possible easiest solution to improve quality of life. Lastly, (Lipsett et al., 2017) proved that exercise during adjuvant radiotherapy for breast cancer has positive impact on reducing fatigue and improve quality of life . However, there are no previous studies to investigate the effect of exercise on trace elements in BC patients nor identifying the optimal dose or parameters of the exercise. So, this study is an attempt to add to the clinical knowledge in this field as it will be the first one that investigates the effect of aerobic exercise on trace elements in women survived BC.

ELIGIBILITY:
Inclusion Criteria:

* All postmenopausal women with breast cancer and received radiotherapy immediately at the end of radiotherapy or max six months to one year in each group. after clinically diagnosed by Oncologist with breast cancer Stage I and II .
* Their ages will range from 50-60 years old.
* Good general Health (ECOG performance status 0-1).
* Voluntary acceptance of participation in the study.

Exclusion Criteria:

* Systematic chronic diseases (respiratory diseases, cardiovascular diseases…etc)
* Cognitive dysfunction as well as neuromuscular or musculoskeletal impairment or disease affecting postural control or motion pattern.
* Professional athletes.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
trace elements levels | 2 months
  blood testing

SECONDARY OUTCOMES:
EORTC QLQ-C30 | 2 months
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Hussein, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided